CLINICAL TRIAL: NCT02540941
Title: Protocols Development for Single Cells Genomics and Their Implementation for Molecular Diversity Between Cells
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 123456- HMO-CTIL
Record Dates: First submitted 2015-06-16; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: non

SUMMARY:
The investigators will extract single cells and analyze the molecular composition of single cells as well as bulks using the latest protocols for single cell and bulk genomics analyses including genetic, epigenetic, transcriptomic and proteomic analyses using the latest available protocols. A broad list of such example protocols are listed below.

The samples and their molecular characterization (including sequencing & molecular levels) will serve as the basis for development of methods for single cells analysis. The developed methods are aimed at genomic transcriptomic, epigenetic, or proteomics analysis of single cells and share the same structure: the measured feature will be translated to a DNA library which will represent the feature by a dedicated assay.

This library alongside with proper mathematical analysis of the sequencing results will be performed in order to conclude the desired feature. The general structure of such protocols is described in our review paper (Single-cell sequencing-based technologies will revolutionize whole-organism science, E. Shapiro, T. Biezuner & S.Linnarsson, Nature Reviews Genetics 14, 618-630, 2013) which is attached to our proposal.

In addition, the researchers will use sequencing based methods (existing and future developed) in order to compare single cells and bulks from different tissues and/or different time points from the same donor in order to measure genetic, epigenetic, transcriptomic, and proteomic diversity.

ELIGIBILITY:
Inclusion Criteria:

Adults

Exclusion Criteria:

* Non

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will obtain human single and bulk cells from healthy donors. Volunteers will be sperm donors who shall designate part or full donation to the proposed research. Egg donors who shall designate part of the eggs to the proposed research; for women who come to the clinics of fertility problems. Reaching the donors will be using advertisements in sperm banks and in women's health centers or asking for student volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Measuring single-cell variability using single-cell genomics | 5 years
  Individual cells samples from multiple tissues, possibly at multiple time points, will be characterized using advanced single-cell genomics protocols. The genomic, transcriptomic and epigenomic signatures of the cells will be measured. Genomic signatures will be used to establish lineage relations among cells. Transcriptomic and epigenomic signatures will be used to characterize cell type and functional state. Statistical analysis will be performed to characterize cell type and state variability and its correlation with lineage relations, tissue of origin and donor age. Bulk samples will be analyzed as controls, as well as for comparing the information gleaned from single-cell analysis to that obtained solely by bulk analysis.